CLINICAL TRIAL: NCT01393834
Title: Delayed Umbilical Cord Clamping Versus Cord Milking in Preterm Neonate - a Randomized, Controlled Trial
Brief Title: Delayed Umbilical Cord Clamping Versus Cord Milking in Preterm Neonate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty with enrollment
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-053
Record Dates: First submitted 2011-06-01; First posted 2011-07-13 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Premature Birth
Keywords: Delayed cord clamping; Umbilical cord; Preterm; Cord milking
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Delayed cord clamping (Experimental): Delayed cord clamping for 30 seconds
  Interventions: Procedure: Delayed cord clamping
- Milking of the cord (Experimental): Milking of the cord 4 times in 10 seconds
  Interventions: Procedure: Milking of the cord
- Immediate cord clamping (No Intervention): Immediate cord clamping after delivery

INTERVENTIONS:
Procedure: Delayed cord clamping — Delay cord clamping for 30 seconds after birth
  Arms: Delayed cord clamping
Procedure: Milking of the cord — Milking of the cord 4 times in 10 seconds
  Arms: Milking of the cord

SUMMARY:
This study is being done to evaluate if delaying cord clamping or milking the umbilical cord of the preterm infant has health benefits for the baby. Timing of clamping of the cord varies among doctors, but there is information that shows that delaying clamping of the umbilical cord in premature infants may reduce the rate of the baby needing a blood transfusion, decrease the risk of infection and bleeding in the head.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or multiples pregnancies in patients admitted for medically indicated delivery or in advanced spontaneous preterm labor with imminent delivery at 24 0/7 - 28 6/7 weeks gestation
* Women ages 18 and older

Exclusion Criteria:

* Planned vaginal breech delivery
* Major fetal abnormalities (defined as those that are lethal or require prenatal or postnatal surgery)
* Fetal death in utero
* Red cell isoimmunization
* Patients who are incapable of informed consent (unconscious, severely ill, mentally handicapped), or are unwilling to undergo randomization
* Placenta previa or other known abnormal placentation (e.g. placenta accreta)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adverse Neonatal Event | up to 24 weeks after birth
  composite of bronchopulmonary dysplasia (BPD), necrotising eneterocolitis (NEC), grade 3 or 4 intraventricular hemorrhage (IVH) or periventricular leukomalacia (PVL), or death prior to discharge home

SECONDARY OUTCOMES:
Maternal estimated blood loss | up to 1 hour after delivery
  Estimated blood loss at delivery
Any grade intraventricular hemorrhage | up to 24 weeks after birth
Severe intraventricular hemorrhage (grade 3 or 4) | up to 24 weeks after birth
Periventricular leukomalacia | up to 24 weeks after birth
Bronchopulmonary dysplasia | up to 24 weeks after birth
Peak transcutaneous and/or serum bilirubin concentrations | up to 24 weeks after birth
Phototherapy | up to 24 weeks after birth
  Requirement and length of phototherapy
Ionotropic support | up to 24 weeks after birth
  Requirement and length of ionotropic support
Neonatal intesive care unit (NICU) length of stay | up to 24 weeks after birth
Sepsis | up to 24 weeks after birth
Necrotizing enterocolitis | up to 24 weeks after birth
Respiratory distress syndrome | up to 24 weeks after birth
Number of blood transfusions while in the neonatal intensive care unit | up to 24 weeks after birth
Ventilator time | up to 24 weeks after birth
Apgar score <7 at 5 minutes | at 5 minutes after birth
Umbilical cord pH < 7.0 | up to 30 minutes after birth
Blood pressure on admission to neonatal intensive care unit | at 30 minutes after birth
Polycythemia | up to 24 hours of life
Hematocrit on admission to neonatal intensive care unit | up to 4 hours after birth
Neonatal death | up to 24 weeks of life
Length of 3rd stage of labor | up to 1 hour after birth
  Time period between delivery of the baby and delivery of the placenta
Use of uterotonic agents | up to 1 hour after birth
Maternal blood transfusion | up to 5 days after delivery
Manual removal of placenta | up to 1 hour after birth
Operating time for cesarean delivery | up to 3 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Rita W Driggers, MD, Principal Investigator — Washington Hospital Center, Georgetown University Hospital